CLINICAL TRIAL: NCT06276179
Title: Epidural Oxycodone for Pain Management for Lower Limb Amputation: A Randomized Controlled Trial
Brief Title: Epidural Oxycodone for Pain Management for Lower Limb Amputation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Gamal Hendawy Shams, Lecturer of Anesthesia and Postsurgical ICU, Faculty of Medicine, Kafrelshiekh University, Kafrelshiekh, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-97
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Epidural; Oxycodone; Pain; Lower Limb Amputation
MeSH Terms: conditions — Pain | interventions — Oxycodone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone (study group) (Experimental): Patient will receive a bolus dose of 0.15 mg/kg plus 20 ml bupivacaine 0.25% followed by an infusion 0.03 mg/kg/h oxycodone plus 0.1 mL/Kg/h bupivacaine 0.125%.
  Interventions: Drug: Oxycodone
- Bupivacaine (control group) (Active Comparator): Patient will receive a bolus 20 ml bupivacaine 0.25% followed by an infusion 0.1 mL/Kg/h bupivacaine 0.125%.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Oxycodone — Patient will receive a bolus dose of 0.15 mg/kg plus 20 ml bupivacaine 0.25% followed by an infusion 0.03 mg/kg/h oxycodone plus 0.1 mL/Kg/h bupivacaine 0.125%.
  Arms: Oxycodone (study group)
Drug: Bupivacaine — Patient will receive a bolus 20 ml bupivacaine 0.25% followed by an infusion 0.1 mL/Kg/h bupivacaine 0.125%.
  Arms: Bupivacaine (control group)

SUMMARY:
The aim of this study is to evaluate the effect of epidural oxycodone for pain management after lower limb amputation.

DETAILED DESCRIPTION:
Phantom limb pain (PLP) is often described as tingling, throbbing, sharp, pins/needles in the limb that is no longer there. It occurs more commonly in upper extremity amputations than lower extremities and tends to be intermittent in frequency. Pain severity varies, and onset can be immediate or years afterward.

The preventive strategies for the PLP pain are difficult to manage and if not addressed adequately may lead to chronic pain. The perioperative role of the anesthesiologist and the acute pain physician is important in the management of somatic and sometimes neuropathic postoperative pain.

Oxycodone is a semi-synthetic narcotic analgesic and historically has been a popular drug of abuse among the narcotic abusing population. Oxycodone is used orally or intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status II or III.
* Undergoing lower limb amputation.
* Under epidural anesthesia.

Exclusion Criteria:

* Hypersensitivity to opioids.
* Cardiac arrhythmias.
* Acute asthma or other obstructive airways disease.
* Severe renal impairment.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain scores | 48 hours postoperatively
  Acute postoperative pain scores will be assessed using numerical rating scale (NRS).Each patient will be instructed about postoperative pain assessment with NRS. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at PACU, 2, 4, 6, 12, 24, 36 and 48 h postoperatively.

SECONDARY OUTCOMES:
Time to the first request for the rescue analgesia | 48 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated). If numerical rating scale (NRS) is more than 3, intravenous morphine 3mg will be administered as rescue analgesia.
Postoperative morphine consumption | 48 hours postoperatively
  Acute postoperative pain scores will be assessed using numerical rating scale (NRS).
  NRS will be assessed at PACU, 2, 4, 6, 12, 24, 36 and 48 h postoperatively. A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. If NRS is more than 3, intravenous morphine 3mg will be administered as rescue analgesia.
Incidence of phantom limb pain | 3 months postoperatively
  Incidence of phantom limb pain will be assessed 3 months after surgery
Adverse effects | 48 hours postoperatively
  Adverse effects such as postoperative nausea and vomiting, pruritus, urinary retention, constipation, and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.